CLINICAL TRIAL: NCT00700245
Title: The Effect of Acute and Chronic Exercise at the Metabolic Syndrome and Markers of Inflammation in Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Tore Christiansen, Department of Medicine and Endocrinology C
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060053
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2008-06-18 (Estimated); Status verified 2008-06

CONDITIONS: Obesity; Healthy
Keywords: Obese; Adults
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- EXO (Active Comparator): Exercise-only (EXO-12 weeks of regular supervised exercise without diet restriction),
  Interventions: Behavioral: Exercise-only (EXO-12 weeks of regular supervised exercise without diet restriction)
- DIO (Active Comparator): Diet-only (DIO-8 weeks of very low energy diet (VLED 600 kcal/d) followed by 4 weeks weight maintenance diet)
  Interventions: Behavioral: Diet-only (DIO-8 weeks of very low energy diet (VLED 600 kcal/d) followed by 4 weeks weight maintenance diet
- DEX (Active Comparator): Diet+exercise (DEX-8 weeks VLED 800 kcal/d + a four weeks weight maintenance diet combined with regular supervised exercise throughout the 12 weeks).
  Interventions: Behavioral: Diet+exercise (DEX-8 weeks VLED 800 kcal/d + a four weeks weight maintenance diet combined with regular supervised exercise throughout the 12 weeks).

INTERVENTIONS:
Behavioral: Exercise-only (EXO-12 weeks of regular supervised exercise without diet restriction) — The exercise intervention for subjects in the EXO consisted of supervised aerobic exercise three times per week with a duration of 60 -75 minutes pr. training session, with an estimated energy expenditure of 500-600 kcal per session. The subjects could choose between different modes of exercise; stationary bicycling, jogging on a treadmill or stair stepping.
  Arms: EXO
Behavioral: Diet-only (DIO-8 weeks of very low energy diet (VLED 600 kcal/d) followed by 4 weeks weight maintenance diet — Subjects in the DIO group were prescribed a liquid VLED(Nupo, Copenhagen) of respectively 600 and 800 kcal pr. day (proteins 41 g, carbohydrates 29 g, fat 5.6 g. pr 100 gram) for eight weeks followed by a weight maintenance diet for four weeks.
  Arms: DIO
Behavioral: Diet+exercise (DEX-8 weeks VLED 800 kcal/d + a four weeks weight maintenance diet combined with regular supervised exercise throughout the 12 weeks). — The exercise intervention for subjects in the DEX group consisted of supervised aerobic exercise three times per week with a duration of 60 -75 minutes pr. training session, with an estimated energy expenditure of 500-600 kcal per session
  Arms: DEX

SUMMARY:
The human adipose and muscle -tissue produce and release a number of bioactive proteins which contributes to the chronic low grade of inflammatory status which is associated with obesity and plays an important role in the pathogenesis of type 2 diabetes and cardiovascular diseases.

Study 1: Our aim is to investigate if exercise has independent and additive effects in combination with diet-induced weight loss on circulating levels of inflammatory markers and mRNA levels in subcutaneous adipose tissue (SAT) and skeletal muscle tissue (SM.

Study 2: Our aim is to investigate whether gender and weight status plays a role in the metabolic response during two hours of acute exercise

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years,
* obese (30 kg/m2 < BMI < 40 kg/m2) physically inactive (<30 minutes pr. day)
* and weight stabile for at least three months (± 2 kg of current body weight)

Exclusion Criteria:

* cardiovascular disease,
* type 2 diabetes, pregnancy or orthopaedic difficulties causing inability to undertake an exercise program

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-06 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Changes in inflammatory markers as Adiponectin, MCP-1, Interleukin-6 and CRP. Moreover changes in body composition quantified with MRI | 8 weeks and 12 weeks
Change in Interleukin-6 and other inflammatory markers in plasma, adipose tissue and muscle tissue | 60, 120 240 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Endocrinology C, Aarhus, Aarhus, Denmark